CLINICAL TRIAL: NCT02632500
Title: Multicenter internAtional raNdomized Controlled manIkin Study on Different Protocols of CPR (MANI-CPR)
Brief Title: Manikin Study on Different Protocols of CPR (MANI-CPR)
Acronym: MANI-CPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pavia nel Cuore (Other)
Collaborators: Robbio nel Cuore (Unknown)
Responsible Party: Principal Investigator, Enrico Baldi, M.D., Pavia nel Cuore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ProtocolsCPR
Record Dates: First submitted 2015-12-10; First posted 2015-12-16 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Quality of Cardio-pulmonary Resuscitation
Keywords: Cardio-Pulmonary Resuscitation; Cardiac Arrest; Training
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 30 compressions and 2 seconds of pause (Experimental): After the randomization the participant will be asked to perform 8 minutes of CPR following the "30 compressions and 2 seconds of pause" protocol (30 chest compressions followed by 2 seconds of pause) on a manikin connected to the Personal Computer.
  Interventions: Other: Quality of chest compressions
- 50 compressions and 5 seconds of pauses (Experimental): After the randomization the participant will be asked to perform 8 minutes of CPR following the "50 compressions and 5 seconds of pause" protocol (50 chest compressions followed by 5 seconds of pause) on a manikin connected to the Personal Computer.
  Interventions: Other: Quality of chest compressions
- 100 compressions and 10 seconds of pause (Experimental): After the randomization the participant will be asked to perform 8 minutes of CPR following the "100 compressions and 10 seconds of pause" protocol (100 chest compressions followed by 10 seconds of pause) on a manikin connected to the Personal Computer.
  Interventions: Other: Quality of chest compressions
- hands-only (Experimental): After the randomization the participant will be asked to perform 8 minutes of CPR following the "hands-only" protocol (continuous chest compressions without any pauses) on a manikin connected to the Personal Computer.
  Interventions: Other: Quality of chest compressions

INTERVENTIONS:
Other: Quality of chest compressions

SUMMARY:
The aim of the study is to verify whether the inclusion of breaks of different frequency and duration during the hands-only cardio-pulmonary resuscitation (CPR) could increase chest compressions quality during an 8-minutes scenario.

DETAILED DESCRIPTION:
Background:

The focus on the hands-only CPR has grown a lot in the last years. The reasons for this are that it's more accepted by lay rescuers, it's easier to remember and to perform, and, above all, it has been demonstrated that it has the same efficacy than standard CPR at least in the first minutes after an out-of-hospital cardiac arrest (OHCA), which are the minutes in which it is more probably that a lay rescuer can intervene. For these reasons ILCOR 2010 and also 2015 guidelines recommended this technique for untrained bystanders or for bystanders who are unwilling to give rescue breaths. ILCOR 2010 and 2015 guidelines have also pointed out that it's not sufficient to perform only a CPR immediately after an OHCA. In fact they have stressed that this CPR must be an high-quality CPR, that is a CPR with compressions of adequate rate (between 100 and 120 per minute) and adequate depth (between 5 and 6 cm), with complete chest recoil between compressions and minimizing interruptions between compressions. This because it has been shown that an high-quality CPR can improve the survival after an OHCA. It has also been demonstrated that the quality of hands-only CPR decades after 1 minute, and considering that the mean time intervention of Emergency Medical System (EMS) on a cardiac arrest scenario in Europe is about 8 minute, it's easy to comprehend that it is very difficult to perform an high-quality CPR with the hands-only technique. It has also been shown that a 10-seconds pause in the hands-only CPR protocol can increase its quality, but, at the moment, there is not a shared protocol to recommend to lay rescuers who are unwilling to give rescue breaths, except to perform chest compressions continuously until EMS arrival.

Purpose:

The aim of the study is to verify whether the inclusion of breaks of different frequency and duration during CPR could increase chest compressions quality during an 8-minutes scenario compared with the hands-only CPR technique.

Materials and Methods:

The study involves multiple training center in Italy and in Europe, that organise Basic Life Support with Automated External Defibrillators (BLS/AED) courses according to ILCOR 2015 guidelines, with an instructor:attendees:manikin ratio of 1:5:1, maximum 1:6:1, and with 1 minute training per participant with real-time feedback using a Laerdal QCPR or Resusci Anne Wireless Skill Reporter manikin connected with a QCPR software. At the end of each course the performance of 1-min of compression-only CPR on the QCPR/Resusci Anne Wireless Skill Reporter manikin without visual feedback for the attendee will be recorded for each participant. In order to eliminate any bias due to heterogeneity of the individual quality of CPR, will be asked to participate in the study to all those who, at the end of this test, will have done the compressions at a rate between 100 and 120 per minute with a result> = 75% in the parameters "percentage of compressions with correct depths (between 5 and 6 cm)", "percentage of correctly released compressions", "percentage of compressions with correct hand position" Those who are between 18 and 80 years old and agree to participate in signing the informed consent, will be randomized to one of four arms of the study. The arms of the study are the 4 different CPR protocols: 30 compressions and 2 seconds of pause (30c2s), 50 compressions and 5 seconds of pause (50c5s), 100 compressions and a 10 seconds of pause (100c10s) and continuous chest compressions without any pauses (hands-only).

The subjects were asked to carry out an 8-minutes performance following the protocol assigned to them on the Laerdal QCPR or Resusci Anne Wireless Skill Reporter manikin connected to the QCPR software without any type of feedback or help.

ELIGIBILITY:
Inclusion Criteria:

* Lay people over 18 years old

Exclusion Criteria:

* Lay people over 80 years old

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-04-28 (Actual); Study Completion 2019-04-28 (Actual)

PRIMARY OUTCOMES:
Chest compressions depth | The whole 8 minutes of the performance carried out by each subject.
  Difference in the percentage of compressions with correct depth (50-60 mm) among the groups

SECONDARY OUTCOMES:
Correctly released compressions | The whole 8 minutes of the performance carried out by each subject.
  Differences in the percentage of correctly released compressions among the groups
Compressions with correct hand position | The whole 8 minutes of the performance carried out by each subject.
  Differences in the percentage of compressions with correct hand position among the groups
Number of compressions per minute | The whole 8 minutes of the performance carried out by each subject.
  Difference in the percentage of compressions with correct rythm among the groups
Pauses to rest | The whole 8 minutes of the performance carried out by each subject.
  Lengths of the pauses taken to rest

CONTACTS AND LOCATIONS:
Locations (8):
- Italy (4):
  - Robbio nel Cuore, Robbio, Pavia
  - Policlinico P. Giaccone, Palermo, PA
  - Centro Studi e Formazione Gymnasium, Pordenone, PN
  - Pavia nel Cuore, Pavia, PV
- Switzerland (4):
  - FormaMed Sàrl, Cortaillod
  - Emergency Training Center, Cugy
  - ES ASUR, Le Mont-sur-Lausanne
  - FCTSA, Lugano

REFERENCES:
- [Derived] Baldi E, Contri E, Burkart R, Borrelli P, Ferraro OE, Paglino M, Pugliesi M, Barbati C, Bertaia D, Tami C, Lopez D, Boldarin S, Denereaz S, Terrapon M, Cortegiani A; and the MANI-CPR investigators. A Multicenter International Randomized Controlled Manikin Study on Different Protocols of Cardiopulmonary Resuscitation for Laypeople: The MANI-CPR Trial. Simul Healthc. 2021 Aug 1;16(4):239-245. doi: 10.1097/SIH.0000000000000505. PMID 32976224
- [Derived] Baldi E, Contri E, Burkart R, Borrelli P, Ferraro OE, Tonani M, Cutuli A, Bertaia D, Iozzo P, Tinguely C, Lopez D, Boldarin S, Deiuri C, Denereaz S, Denereaz Y, Terrapon M, Tami C, Cereda C, Somaschini A, Cornara S, Cortegiani A. Protocol of a Multicenter International Randomized Controlled Manikin Study on Different Protocols of Cardiopulmonary Resuscitation for laypeople (MANI-CPR). BMJ Open. 2018 Apr 19;8(4):e019723. doi: 10.1136/bmjopen-2017-019723. PMID 29674365